CLINICAL TRIAL: NCT03624959
Title: A Phase 1, Randomized, Parallel-Group, Open-Label Study to Evaluate the Effect of the Modulators of the Cytochrome P450 (CYP) 2C8 and/or 3A on the Single-Dose Pharmacokinetics of Ozanimod and CC112273 in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of Ozanimod With Inhibitor or Inducer of CYP2C8 and/or CYP3A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RPC01-1912; U1111-1215-6965 (Other: WHO)
Record Dates: First submitted 2018-07-06; First posted 2018-08-10 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Cytochrome P450 (CYP); ozanimod
MeSH Terms: interventions — ozanimod; Gemfibrozil; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment Group A - Ozanimod 0.46mg (Experimental): A single dose of ozanimod 0.46 mg on Day 1
  Interventions: Drug: Ozanimod
- Treatment Group B - Ozanimod plus Gemfibrozil (Experimental): Gemfibrozil 600 mg twice daily (BID) on Days 1 through 17. On Day 4, a single dose of ozanimod 0.46 mg will be coadministered with the morning dose of gemfibrozil.
  Interventions: Drug: Ozanimod; Drug: Gemfibrozil
- Treatment Group C - Ozanimod 0.92mg (Experimental): A single dose of ozanimod 0.92 mg on Day 1.
  Interventions: Drug: Ozanimod
- Treatment Group D - Ozanimod plus Itraconazole (Experimental): Itraconazole 200 mg once daily (QD) on Days 1 through 17. On Day 4, a single dose of ozanimod 0.92 mg will be co-administered with itraconazole.
  Interventions: Drug: Ozanimod; Drug: Itraconazole
- Treatment Group E - Ozanimod plus Rifampin (Experimental): Rifampin 600 mg QD on Days 1 through 21. On Day 8, a single dose of ozanimod 0.92 mg will be coadministered with rifampin
  Interventions: Drug: Ozanimod; Drug: Rifampin

INTERVENTIONS:
Drug: Ozanimod — ozanimod
Drug: Gemfibrozil — Gemfibrozil
  Arms: Treatment Group B - Ozanimod plus Gemfibrozil
Drug: Itraconazole — Itraconazole
  Arms: Treatment Group D - Ozanimod plus Itraconazole
Drug: Rifampin — Rifampin
  Arms: Treatment Group E - Ozanimod plus Rifampin

SUMMARY:
The purpose of this study is to evaluate the effect of the following index inhibitors or inducers of CYP2C8 and/or CYP3A on the single-dose pharmacokinetics (PK) of ozanimod and its major active metabolite, CC112273, in healthy adult subjects: gemfibrozil (strong inhibitor of CYP2C8), rifampin (moderate inducer of CYP2C8 and strong inducer of CYP3A), and itraconazole (strong inhibitor of CYP3A).

Study Design

This is a Phase 1, randomized, parallel-group, open-label study with two parts, 1 and 2. Forty subjects will be enrolled in Part 1 and will be randomized into 1 of the 2 treatment groups, with 20 subjects in each treatment group. Sixty subjects will be enrolled in Part 2 and will be randomized into 1 of the 3 treatment groups, with 20 subjects in each treatment group. . Study parts and treatment groups are as follow:

Part 1:

* Treatment Group A (reference): A single dose of ozanimod.
* Treatment Group B (test): Gemfibrozil 600 mg twice daily (BID) on Days 1 through 17. On Day 4, a single dose of ozanimod will be coadministered with the morning dose of gemfibrozil.

Part 2:

* Treatment Group C (reference): A single dose of ozanimod.
* Treatment Group D (test): Itraconazole 200 mg once daily (QD) on Days 1 through 17. On Day 4, a single dose of ozanimod will be coadministered with itraconazole.
* Treatment Group E (test): Rifampin 600 mg QD on Days 1 through 21. On Day 8, a single dose of ozanimod will be coadministered with rifampin.

Study Population Subjects will be healthy men and non-pregnant, non-lactating women, ages 18 to 55 years, inclusive, with a body weight of at least 110 pounds (50 kg); body mass index (BMI) within the range of 18.0 to 30.0 kg/m2, inclusive.

Length of Study The study duration ranges from 43 days to 50 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a man or non-pregnant, non-lactating woman, ages 18 to 55 years, inclusive, at the time of signing of the informed consent form (ICF).
2. Female subjects must meet at least 1 of the following criteria:

   * Negative serum pregnancy test at Screening and Day -1 (women of child-bearing potential [WOCBP] only).
   * Postmenopausal (defined as 2 years after the last period and follicle-stimulating hormone [FSH] > 40 IU/L).
   * Received surgical sterilization (eg, bilateral tubal ligation, bilateral oophorectomy, hysterectomy) at least 6 months before Screening with medical records.
3. Females of child-bearing potential:

   Must agree to practice a highly effective method of contraception throughout the study until completion of the 75-day Safety Follow-up. Highly effective methods of contraception are those that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly.

   Acceptable methods of birth control in this study are the following:
   * Combined hormonal (oestrogen and progestogen containing) contraception, which may be oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, implantable
   * Placement of an intrauterine device or intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Sexual abstinence

   Male subjects:

   Must agree to use a latex condom with spermicide during sexual contact with WOCBP while participating in the study and until completion of the 75-day Safety Follow-up.

   All subjects:

   Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception. Female condom and male condom should not be used together.
4. Male subjects must agree to refrain from donating sperm throughout the study and until completion of the 75-day Safety Follow-up.
5. Subject has a body weight of at least 110 pounds (50 kg); body mass index (BMI) within the range of 18.0 to 30.0 kg/m2, inclusive (Screening and Day -1).
6. Subject is in good health, as determined by no clinically significant findings from medical or surgical history, 12-lead ECG, physical examination, clinical laboratory tests, and vital signs.
7. Subject must be able to comprehend and provide written informed consent, and must be able to comply with the requirements of the study, including the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Subject with a seated blood pressure outside 90 to 140 mmHg systolic or 50 to 90 mmHg diastolic at Screening or Day -1.
2. Subject with a seated pulse rate outside 55 to 90 bpm at Screening or Day -1.
3. Subject has a presence or history of any abnormality or illness that, in the opinion of the investigator, may affect absorption, distribution, metabolism, or elimination of the Investigational product (IP) or would limit the subject's ability to participate in and complete this clinical study.
4. Subject has a history of alcoholism, drug abuse, or addiction within 24 months prior to Screening.
5. Subject has a positive serum test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
6. Subject has used any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, electronic cigarettes, vape, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) or marijuana (cigarette, joint, vape, edibles, etc) within 3 months prior to the first dose of IP.
7. Subject has a positive urine drug test including cotinine at Screening or Day -1.
8. Subject has a positive alcohol urine or breath test at Screening or Day -1.
9. Subject has received any investigational drug within 30 days or 5 times the elimination half-life (if known), whichever is longer, prior to the first dose of IP.
10. Subject has used any systemic over-the-counter medication (excluding acetaminophen up to 1 g/day), dietary or herbal supplement (excluding vitamins/multivitamins) within 7 days prior to the first dose of IP. St. John's wort, naringenin, curcurmin/turmeric, passion flower, and quercetin must be discontinued at least 28 days prior to the first dose of IP.
11. Subject has used any systemic prescription medication (excluding hormonal contraceptives) within 28 days or 5 times the elimination half-life, whichever is longer, prior to the first dose of IP.
12. Subject has ingested alcohol within 7 days prior to the first dose of IP.
13. Subject fails or is unwilling to abstain from strenuous physical activities for at least 24 hours prior to the first dose of IP.
14. Subject has poor peripheral venous access.
15. Subject has donated greater than 400 mL of blood within 60 days prior to Day 1.
16. Subject has a history of any medical condition or medical history that, in the opinion of the investigator, might confound the results of the study or jeopardize the safety or welfare of the subject.
17. Subject has history of hypersensitivity or allergic reaction to S1P receptor modulators (both Parts 1 and 2), gemfibrozil (Part 1 only), itraconazole or other azole antifungals (Part 2 only), or rifampin (Part 2 only).
18. Subject has a history of gall bladder disease (Part 2 only).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics- Cmax | Up to 14 days after ozanimod dosing
  Maximum observed plasma concentration
Pharmacokinetics- AUC∞ | Up to 14 days after ozanimod dosing
  Area under the concentration-time curve from time 0 to infinity
Pharmacokinetics- AUC0-14d | Up to 14 days after ozanimod dosing
  Area under the concentration-time curve from time 0 to 14 days post dose

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 75 days after ozanimod dosing
  The incidence, severity, and relationship of TEAEs
Pharmacokinetics- Tmax | Up to 14 days after ozanimod dosing
  Time to Cmax
Pharmacokinetics- CL/F | Up to 14 days after ozanimod dosing
  Apparent oral clearance
Pharmacokinetics- Vz/F | Up to 14 days after ozanimod dosing
  Apparent volume of distribution during terminal phase after oral administration
Pharmacokinetics- λz | Up to 14 days after ozanimod dosing
  Terminal elimination rate constant
Pharmacokinetics- t1/2 | Up to 14 days after ozanimod dosing
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tran, Pharm.D, Study Director — Celgene Corporation
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

REFERENCES:
- [Derived] Tran JQ, Zhang P, Ghosh A, Liu L, Syto M, Wang X, Palmisano M. Single-Dose Pharmacokinetics of Ozanimod and its Major Active Metabolites Alone and in Combination with Gemfibrozil, Itraconazole, or Rifampin in Healthy Subjects: A Randomized, Parallel-Group, Open-Label Study. Adv Ther. 2020 Oct;37(10):4381-4395. doi: 10.1007/s12325-020-01473-0. Epub 2020 Aug 28. PMID 32857315